CLINICAL TRIAL: NCT04393181
Title: IMPact of Donor Heart Function on Recipient Outcomes - a prospectiVE Study to Increase the Utilization of Donor HEARTs
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: IMPROVED HEART
Record Dates: First submitted 2020-05-13; First posted 2020-05-19 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Heart Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — The hearts of organ donors that are not transplanted will be used for tissue analysis when logistically feasible and permission is granted, in accordance with current regulations. The hearts will be examined for coronary heart disease and heart attack. Tissue samples will be taken from several areas with affected (in such donors) or normal function.
  Blood samples from donors will be taken when logistically feasible and permission is granted, in accordance with current regulations.
  From the donors, 20 ml blood is planned to be taken on up to three occasions, i.e. a total of 60 ml blood. Blood samples for analysis of troponin T and NTproBNP will be taken as part of normal healthcare routines and destroyed immediately after analysis .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- recipients of hearts with impaired function: Patient who has been accepted for heart transplantation at the participating transplantation center and who will receive heart with impaired function
  Interventions: Procedure: Heart transplantation 1
- recipients of hearts with normal function: Patient who has been accepted for heart transplantation at the participating transplantation center and who will receive heart with normal function
  Interventions: Procedure: Heart transplantation 2

INTERVENTIONS:
Procedure: Heart transplantation 1 — Heart transplantation will be performed according to local routines. Recipients will be transplanted with a donor heart with left ventricular dysfunction, defined as an ejection fraction less than 50% or regional hypokinesia.
  Groups: recipients of hearts with impaired function
Procedure: Heart transplantation 2 — Heart transplantation will be performed according to local routines. Recipients will be transplanted with a donor heart with normal function, according to the recommendations from The International Society for Heart and Lung Transplantation (ISHLT).
  Groups: recipients of hearts with normal function

SUMMARY:
Severe heart failure is a diagnosis with a very poor prognosis. Heart transplantation is the best treatment for terminal heart failure but this type of treatment is limited by the number of available organs. About 20-25% of possible donor hearts are not considered for transplantation because they have some form of functional impairment. The functional impairment affecting organ donors is, however, usually reversible. A number of retrospective studies show that cardiac function recovers and recipients of hearts with dysfunction do not have worse outcomes compared to recipients of hearts with perfect cardiac function. However, there are no prospective studies on whether the functional impairment of the donor heart is of significance for the recipient. With a systematic and simple investigation of the heart, it should be possible to identify the hearts that are safe to transplant. This will thus increase the number of available donors.

DETAILED DESCRIPTION:
Severe heart failure is a diagnosis with a very poor prognosis where the 2-year mortality rate for serious heart failure is over 50%, which exceeds many cancer diagnoses. Despite advances in pharmacological treatment and mechanical pumps, heart transplantation is considered to be the best treatment for terminal heart failure. However, heart transplantation as a treatment for terminal heart failure is limited by the number of available organs. If the investigators could take care of more organs, more patients could be transplanted. It is therefore of the utmost importance that every heart that can be transplanted successfully is considered.

According to current recommendations, a heart should be in near perfect condition to be considered for transplantation. For a donor heart to be transplanted, it should not exhibit:

* More than mild-to-moderate cardiac impairment (EF < 40%)
* Regional discrete wall motion abnormalities
* Need for excessive inotropic support (dobutamine >20µg/kg/minute)
* Intractable ventricular arrhythmias.

Cardiac dysfunction in organ donors, however, is usually secondary to the disease that led to brain death and is reversible; there is nothing wrong with the heart itself but it has ended up in an unfavorable environment that temporarily affects its function. A common cause of cardiac dysfunction in organ donors is stress-induced cardiomyopathy/Takotsubo cardiomyopathy. Stress-induced cardiomyopathy is a relatively newly described acute cardiac syndrome in which the heart develops regional wall motion abnormalities caused by severe catecholamine stimulation of the myocardium. In the organ donor, a strong catecholamine storm is observed in combination with compression and the development of brain death, which can trigger stress-induced cardiomyopathy. This type of change is seen in 20-25% of potential organ donors. One of the most important characteristics of stress-induced cardiomyopathy is its rapid recovery, however, and cardiac function is usually normalized within a few hours or Days 8-10. This is not only seen as a functional recovery, but also a structural and biochemical recovery of the heart. In addition to organ donors with intracranial events, stress-induced cardiomyopathy is also seen in patients with hypoxic/anoxic brain injuries as a result of hypoxic cardiac arrest, and even in these cases, cardiac events are temporary.

There are potentially differential diagnoses for stress-induced cardiomyopathy in potential donors. The most important is ischemic heart disease which can quickly and relatively easily be diagnosed with coronary angiography. Coronary angiography is performed today on approximately one-third of potential donors and then primarily on donors with a risk profile for coronary artery disease. Another different diagnosis is myocarditis, which does not have the same reversibility as stress-induced cardiomyopathy and usually gives a different echocardiographic image.

The recommendation not to utilize hearts with regional wall motion abnormalities has inadequate scientific support. The recommendation is based on a retrospective study that is over 30 years old and did not have cardiac dysfunction as the primary outcome measure. Upon review of this article, the data does not support the idea that regional wall motion abnormalities would be associated with worse outcomes. Despite this, this recommendation has been the basis for deciding whether to transplant the heart or not. There is a wariness, especially with American thoracic surgeons, to take into account such hearts. There is a number of retrospective studies that show that the outcome is not worse for patients who have been transplanted with hears that have/have had dysfunction. The main studies are presented below:

* A study based on material from the USA (UNOS database) in which patients who received a heart with ejection fraction <50% (n=740) were identified and compared with recipients of hearts with normal function (n=30253). No difference in mortality at one year after transplantation was observed between the groups.
* A study based on the same material showed that long-term survival was not inferior for recipients of hearts with ejection fraction<50%. Cardiac function was also the same for recipients of hearts with normal function and impaired function one year after transplantation.
* In a study based on the same database (UNOS database) 472 recipients who received a heart with improved function, defined as EF≤40% at one examination and EF≥50% at a follow-up examination, were identified. The control group were recipients of hearts with normal function EF≥55%. There was no difference in mortality, primary graft failure, allograft vasculopathy between the groups, even when propensity score matching was applied.
* A study based on other material from the USA (California Transplant Donor Network) reported figures where low ejection fraction (EF<50%, number of patients not reported) or regional hypokinesia (n=197) did not affect outcome.
* An older study based on material from the USA showed that regional hypokinesia has no bearing on recipients' mortality. The number of patients with regional hypokinesia was not reported but 1719 patients were included in the study.
* A study from Transplantation Centre, Sahlgrenska, analyzed donors and recipients during a 10-year period. In total, 641 donors were included in the analyses and 155 (24%) of the donors had cardiac dysfunction. Recipients of hearts with dysfunction (n=42) did not have worse outcomes (death, retransplantation) compared to recipients of hearts with normal function. Short-term outcomes (intensive care unit (ICU) care time, advanced hemodynamic support, postoperative dialysis, rejection) also did not differ between the groups. Cardiac function was rapidly recovered in the recipients and both groups had the same ejection fraction already a few days after transplantation.

These retrospective studies form a relatively good foundation and cover almost 1400 patients. However, prospective studies on transplantation of hearts with functional impairment are missing.

At Transplantation Centre, Sahlgrenska, there are many years of experience of handling hearts with impaired function. This clinical experience suggests that it is not associated with complications. The studies referenced above confirm this experience.

Overall, there is room to increase the number of heart donors, and thus the number of heart transplantations, if the heart donors with reversible dysfunction are utilized. This study aims to prospectively investigate the cardiac function of donors and evaluate if it is of significance to the outcome of the recipient. The study sets guidelines for investigative procedures as well as which hearts should be transplanted, based on previous retrospective studies. The investigators expect that the recipients' outcome will not be affected by the cardiac function of the donor, provided the study's recommendations are followed. Our data shows that approximately every fourth potential heart donor suffers from functional impairment. This is in line with other studies that observed that about 20% of hearts are refused due to affected function. The investigators estimate that a systematic consideration of these hearts can increase the number of transplantations by 20-30%.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has been accepted for heart transplantation at the participating transplantation center

  * The research subject has given written consent to participate in the study
  * Aged 18 years or older

Exclusion Criteria:

* • Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation

  * Another study, where the patient is included, which is not considered compatible with the current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with severe heart failure accepted for heart transplantation at Transplantationscentrum, Sahlgrenska University Hospital, Gothenburg, Sweden
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Dead | One year after heart transplantation.
  Death, retransplantation or need of a mechanical heart pump.

SECONDARY OUTCOMES:
Frequency | 24 hour after transplantation
  Frequency of left-sided moderate or severe primary graft dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Göran Dellgren, MD, PhD, Principal Investigator — Vastragotalandsregionen, Sahlgrenska University Hospital,Gothenburg, Sweden
Locations (1):
- Sahlgrenska University Hostpial, Gothenburg, Västra Götaland County, Sweden